CLINICAL TRIAL: NCT01006902
Title: Outcomes of Oncology Therapy in the Elderly: Trajectory of Functional Decline and Correlates of Change
Status: Terminated | Type: Observational
Why Stopped: Insufficient recruitment
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Kim Dittus, MD, PhD, Assistant Professor, University of Vermont
Other Study IDs: Oncology therapy in elderly
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Cancer
Keywords: Elderly; Function; Oncologic therapy; Functional change with chemotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples will be obtained and stored at -80 degrees celsius
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Individuals age 65 or older: Individuals age 65 or older receiving chemotherapy for cancer or short term androgen deprivation therapy for individuals 65 or older with prostate cancer.

SUMMARY:
The proposed project will document the degree of function decline, assess the relationship between function and cancer- related symptoms and evaluate relationships between function and quality of life. Participants are evaluated before therapy, after therapy and again 3 months post therapy to evaluate functional change. Knowledge gained will help us plan interventions around the time of cancer therapy to help older adults preserve or improve function.

DETAILED DESCRIPTION:
The study looks at functional change of elderly cancer patients. Approximately 52 cancer patients age 65 or older will be asked to participate. Cancer patients asked to participate will be receiving cancer therapy with the intention of providing a cure. Functional change will be assessed from the time of diagnosis, through therapy to the early post therapy time frame. A comprehensive model explaining reasons for function change is used as the framework for choosing variables to measure. Components of function that will be measured include a 6 minute walk test, lower extremity muscle strength, a Short Physical Performance Battery assessing function of legs and a test that simulates typical household activities. Surveys will be used to subjects own assessment of their activity and function. The four most common cancer-related side effects will be measured and include fatigue, sleep impairment, shortness of breath and pain. Some markers in the blood may be abnormal and be related to declines in function. They will also be measured. Differences in function over time will be determined and relationships between function, cancer-related side effects and quality of life will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older
* Diagnosis of a malignancy requiring chemotherapy as part of intent to cure oncologic therapy or diagnosis of prostate cancer requiring 6 months or less of androgen deprivation therapy as part of oncologic treatment.
* A planned oncologic regimen of at least 3 months but not more than 9 months excluding surgery. This will include most solid tumors and lymphoma.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior treatment for malignancy other than basal or squamous cell skin cancer
* Evidence of metastatic disease
* Individuals with acute and chronic leukemias and individuals receiving anti-estrogen therapy only as their primary oncologic treatment.
* Dementia, psychotic condition or other central nervous system impairment limiting compliance
* Medical conditions that limit ability to walk at least 4 meters.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Individuals age 65 or older diagnosed with a malignancy and receiving chemotherapy or androgen deprivation therapy as part of their oncology therapy.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2009-11; Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Determine change from baseline of physical function in elderly cancer patients after oncologic therapy. | Baseline, post therapy, 3 months post therapy
Identify the relationship between cancer-related symptoms and physical function during oncologic therapy | at end of therapy

SECONDARY OUTCOMES:
Measure changes in quality of life during and after oncologic therapy | Baseline, post therapy, 3 months post therapy
Evaluate the relationship between functional status and quality of life in elderly cancer patients receiving oncologic therapy | Baseline, post therapy, 3 months post therapy

CONTACTS AND LOCATIONS:
Overall Officials: Dittus Kim, MD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont/Fletcher Allen Health Care, Burlington, Vermont, United States